CLINICAL TRIAL: NCT04512066
Title: A Phase II, Multi-Center, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Trial of the Efficacy and the Safety of RO6889450 (Ralmitaront) vs Placebo in Patients With an Acute Exacerbation of Schizophrenia or Schizoaffective Disorder
Brief Title: A Trial of the Efficacy and the Safety of RO6889450 (Ralmitaront) vs Placebo in Patients With an Acute Exacerbation of Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP41743
Record Dates: First submitted 2020-08-12; First posted 2020-08-13 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia, Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 150 mg Once Daily (QD) RO6889450 (Experimental): Participants will receive 150 mg of RO6889450 QD for 4 weeks or 12 weeks or 48 weeks.
  Interventions: Drug: RO6889450
- 45 mg QD RO6889450 (Experimental): Participants will receive 45 mg of RO6889450 QD for 4 weeks or 12 weeks or 48 weeks.
  Interventions: Drug: RO6889450
- Placebo (Placebo Comparator): Participants will receive oral placebo QD for 4 weeks. Participants from this arm that continue to the extension period will be randomized to either 45 mg or 150 mg QD of RO6889450 for up to an additional 8 weeks or additional 44 weeks (optional 36-Week Safety Extension Phase).
  Interventions: Drug: Placebo
- 4 mg QD Risperidone (Active Comparator): Participants will receive 4 mg of risperidone QD for 4 weeks or 12 weeks or 48 weeks.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: RO6889450 — Participants will receive oral RO6889450 QD.
  Arms: 150 mg Once Daily (QD) RO6889450; 45 mg QD RO6889450
Drug: Placebo — Participants will receive oral placebo QD.
  Arms: Placebo
Drug: Risperidone — Participants will receive oral risperidone QD.
  Arms: 4 mg QD Risperidone

SUMMARY:
This study will investigate the efficacy and safety of RO6889450 as monotherapy in participants experiencing an acute exacerbation of symptoms of schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion criteria

* Participant must be 18 to 45 years of age inclusive
* Participants with a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of schizophrenia or schizoaffective disorder as confirmed by the Mini International Neuropsychiatric Interview (MINI)
* Disease duration </=10 years
* Have a current acute exacerbation of schizophrenia of no more than 8 weeks before screening visit and no current signs of apparent lack of treatment response
* At the time of screening, the participant needs to be either hospitalized or requiring inpatient psychiatric care according to clinical judgment. If the participant has been hospitalized for the current exacerbation, the hospitalization has to be of a maximum of 1 week prior to screening.
* In previous exacerbations and hospitalizations, the subject has shown a pattern of response to appropriate antipsychotic treatment
* Medically stable over a period of 3 months (non-psychiatric conditions) prior to screening visit and not expected to require hospitalization or change of treatment for non-psychiatric conditions for the duration of the study
* Screening and baseline CGI-S >/=4 (moderate or worse)
* Screening and baseline PANSS total score >= 80
* Based on screening and baseline PANSS, scores of >/= 4 (moderate or worse) on 2 or more of the following items: delusions, conceptual disorganization, unusual thought content, hallucinatory behavior, or suspiciousness/persecution
* Body mass index between 18 and 35 kg/m2 inclusive
* Male and female participants; female participants agree to remain abstinent or use acceptable contraceptive methods during the treatment period and for at least 28 days after the last dose of study drug

Additional inclusion criteria for optional 36-Week Safety Extension Phase

* Successful completion of the 12-week treatment period
* No signs or symptoms of worsening of the psychiatric or medical status that would preclude the patient from the participation in the 36-Week Safety Extension Phase or affect their ability to comply with the study requirements.

Exclusion criteria

* Has been inpatient for > 1 week or had any other hospitalization for acute exacerbation of schizophrenia or schizoaffective disorder within the prior 8 weeks or signs of lack of response to antipsychotic treatment
* Disease duration > 10 years
* Is currently an inpatient on an involuntary basis
* Subject answers "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) or any suicidal behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS) assessment within one month from screening or between screening and baseline
* Lifetime history of homicidal behavior
* Moderate to severe substance use disorder within six months (excluding nicotine) as defined by DSM-5
* Other current DSM-5 diagnosis (e.g., bipolar disorder, major depressive disorder)
* A prior or current general medical condition that might be impairing cognition or other psychiatric functioning (e.g., migraine headaches requiring prophylaxis treatment, head trauma, dementia, seizure disorder, stroke; or neurodegenerative, inflammatory, infectious, neoplastic, toxic, metabolic, or endocrine conditions)
* Clinically significant abnormalities in laboratory safety test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis), including a) Aspartate aminotransferase (AST), OR alanine aminotransferase (ALT) 2 x upper limit of normal (ULN), OR total bilirubin > 1.5 ULN with the exception of known Gilbert syndrome. b) Serum creatinine > 1.5 ULN
* Positive result at screening for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV, untreated), or human immunodeficiency virus (HIV)-1 and -2. HCV participants who have been successfully treated and who test negative for HCV RNA are eligible for entry into the study
* Tardive dyskinesia that is moderate to severe or requires treatment
* History of neuroleptic malignant syndrome
* Average triplicate QTcF interval greater than 450 msec for males and 470 msec for females or other clinically significant abnormality on screening ECG based on centralized reading
* Participant for whom risperidone is contraindicated or who have a documented history of lack of response or intolerance to risperidone or paliperidone or participants with known hypersensitivity to risperidone, paliperidone, or to any excipients in Risperdal
* Participant treated with a long acting injectable antipsychotic or other antipsychotics that cannot be washed-out within the allotted screening period
* History of electro-convulsive therapy (ECT) for any reason
* Participant treated with clozapine at any dose within 12 months of screening visit or participants treated with clozapine at 200 mg/day or above at any time; low dose (< 200mg/day) use for insomnia or dyskinesia longer than 12 months prior to screening visit is permitted
* Participants currently receiving a psychotropic or other medication used as a psychotropic, which cannot be discontinued during the screening period
* Positive urine drug screen for amphetamines, methamphetamines, opiates, buprenorphine, methadone, cocaine and barbiturates. In case of positive urine drug screen for cannabinoids, the participant may be allowed to enter the study if approved by Medical Monitor
* Participant has previously received RO6889450
* Participant received an investigational drug within 28 days or five times the half-life of the investigational drug prior to the first study drug administration
* Diagnosis of COVID-19 infection (confirmed or presumptive) 4 weeks prior to screening or during screening. Participants can be re-screened after 4 weeks of full recovery in addition to investigator and/or institutional approval to enroll

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 287 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (24):
  - Woodland International Research Group Inc., Little Rock, Arkansas
  - CITrials, Inc., Bellflower, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - California Clinical Trials Medical Group managed by Parexel, Glendale, California
  - Synergy San Diego, Lemon Grove, California
  - NRC Research Institute, Orange, California
  - ASCLEPES Research Centers, Panorama City, California
  - CNRI - Los Angeles, LLC, Pico Rivera, California
  - CITrials, Inc., Riverside, California
  - California Neuropsychopharmacology Clinical Research Institute, LLC, San Diego, California
  - Artemis Institute For Clinical Research LLC - San Diego - ClinEdge - PPDS, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Galiz Research, LLC, Hialeah, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Premier Clinical Research Institute - Miami - BTC - PPDS, Miami, Florida
  - Research Centers of America - ERG, Oakland Park, Florida
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - CBH Health LLC, Gaithersburg, Maryland
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Midwest Clinical Research Center - ERG - PPDS, Dayton, Ohio
  - Community Clinical Research Inc., Austin, Texas
  - Pillar Clinical Research LLC, Garland, Texas
- Japan (2):
  - National Center of Neurology and Psychiatry, Tokyo
  - Seishinkai Okehazama Hospital Fujita Kokoro Care Center, Toyoake
- Russia (8):
  - Psychiatry Hospital #1 n.a. P.P.Kashchenko, Saint Petersburg, Sankt-Peterburg
  - Leningradskiy Regional Psychoneurologic Dispensary, Saint Petersburg, Sankt-Peterburg
  - Psychiatric Hospital St Nicholas the Wonderworker, Saint Petersburg, Sankt-Peterburg
  - City Psychiatry Hospital #3 n.a. I.I. Skvortsov-Stepanov, Saint Petersburg, Sankt-Peterburg
  - FSBI National Medical Research Centre of Psychiatry and Neurology n.a. V.M. Bekhterev of MoH of RF, Sankt-peterburg, Vladimirskaya Oblast’
  - Saratov regional clinical psychoneurological hospital St Sofii, Saratov
  - Stavropol Regional Psychiatry Hospital #2, Stavropol
  - Tomsk National Scientific Medical Center of Russian Academy of Sciences, Tomsk
- Ukraine (6):
  - Communal Non-Commercial Enterprise of Kharkiv RC Regional clinical psychiatric hospital #3, Kharkiv, Kharkiv Governorate
  - Public NPE Kherson Regional Institution of Mental Care of Kherson RC, Kherson, Kherson Governorate
  - Kyiv Medical Regional Union Psychiatry, Kylv, KIEV Governorate
  - Communal Non-Commercial Enterprise Cherkasy Regional Psychiatric Hospital of Cherkasy RC, Smila, KIEV Governorate
  - Communal NPE Vinnytsia Reg. Clin. Psychoneurolog. Hosp. n.a. O.I. Yushchenko of Vinnytsia RC, Vinnytsia, Podolia Governorate
  - Poltava Regional Psychiatry Hospital, Poltava, Poltava Governorate

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Halff EF, Rutigliano G, Garcia-Hidalgo A, Howes OD. Trace amine-associated receptor 1 (TAAR1) agonism as a new treatment strategy for schizophrenia and related disorders. Trends Neurosci. 2023 Jan;46(1):60-74. doi: 10.1016/j.tins.2022.10.010. Epub 2022 Nov 8. PMID 36369028

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 287 participants initially randomized in the double-blind treatment period. 11 excluded from final analysis due to having not received assigned study medication or because of re-enrollment. Participants were not required to participate in all study parts and those that did not continue to the double-blind treatment period either discontinued the study during the double-blind treatment period or exited the study after completing the period. 197 continued to the double-blind extension period.
Groups:
- Placebo: Participants received oral placebo QD for 4 weeks. Participants from this arm that continued on to the extension period were randomized to either 45 mg or 150 mg QD of RO6889450 for up to an additional 8 weeks, or up to an additional 44 weeks if they continued to the optional 36-week safety extension.
  Note: This arm was only in the double-blind treatment period.
- RO6889450 45 mg: Participants received 45 mg of RO6889450 QD for 4, 12, or 48 weeks.
- RO6889450 150 mg: Participants received 150 mg of RO6889450 QD for 4, 12, or 48 weeks.
- Risperidone 4 mg: Participants received 4 mg of risperidone QD for 4, 12, or 48 weeks.
- Placebo - RO6889450 45 mg: Participants from the placebo arm in the double-blind treatment period that continued on to the extension period were randomized to either 45 mg or 150 mg once daily (QD) of RO6889450 for up to an additional 8 weeks, or up to an additional 44 weeks if they continued to the optional 36-week safety extension.
  Note: This arm started in the extension period.
- Placebo - RO6889450 150 mg: Participants from the placebo arm in the double-blind treatment period that continued on to the extension period were randomized to either 45 mg or 150 mg QD of RO6889450 for up to an additional 8 weeks, or up to an additional 44 weeks if they continued to the optional 36-week safety extension.
  Note: This arm started in the extension period.
Period: Double-blind Treatment Period
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg | Placebo - RO6889450 45 mg | Placebo - RO6889450 150 mg
Started | 73 | 71 | 69 | 74 | 0 | 0
Completed | 56 | 55 | 53 | 60 | 0 | 0
Not Completed | 17 | 16 | 16 | 14 | 0 | 0
Not completed — Adverse Event | 6 | 4 | 5 | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 3 | 5 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 9 | 5 | 12 | 0 | 0
Period: Extension Period
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg | Placebo - RO6889450 45 mg | Placebo - RO6889450 150 mg
Started | 0 | 44 | 46 | 56 | 25 | 26
Completed | 0 | 30 | 26 | 38 | 9 | 12
Not Completed | 0 | 14 | 20 | 18 | 16 | 14
Not completed — Adverse Event | 0 | 1 | 4 | 3 | 1 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 4 | 4 | 1 | 3 | 3
Not completed — Lost to Follow-up | 0 | 1 | 5 | 2 | 3 | 2
Not completed — Non-compliance with study drug | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 7 | 11 | 8 | 4

BASELINE CHARACTERISTICS:
Population: The efficacy analysis population (EAP) was used to determine baseline characteristics. The EAP included all randomized participants who received at least one dose of study medication and who had primary efficacy assessments at baseline and on at least one occasion post-baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg | Total
Number analyzed (Participants) | 72 | 65 | 68 | 71 | 276
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.2 (7.1) | 34.0 (7.0) | 32.3 (6.5) | 32.9 (7.1) | 33.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 15 | 18 | 71
  Male | 53 | 46 | 53 | 53 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 8 | 10 | 37
  Not Hispanic or Latino | 64 | 54 | 60 | 61 | 239
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 33 | 27 | 32 | 31 | 123
  White | 37 | 35 | 32 | 39 | 143
  More than one race | 0 | 1 | 2 | 0 | 3
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 4
Description: The PANSS is a 30-item rating scale that evaluates positive, negative, and other symptoms in patients with schizophrenia. The Positive subscale is a 7-item scale that assesses features in schizophrenia that are not present in a normal mental state. The Negative subscale is a 7-item scale that assesses features absent in schizophrenia but present in those with a normal mental state. Items are rated on a 7-point scale, where 1 = absent and 7 = extreme, for a maximum score of 49 for each scale. The General subscale is a 16-item scale that assesses the overall severity of schizophrenia and the risk of aggression. Items are rated on the same scale, with a minimum score of 16 and a maximum score of 112. Total scores are calculated by adding subscale scores together, for a minimum score of 30 and a maximum score of 210. Higher scores indicate higher severity.
Time Frame: Week 4 (Day 28)
Population: The efficacy analysis population (EAP) included all randomized participants who received at least one dose of study medication and who had primary efficacy assessments at baseline and on at least one occasion post-baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 72 | 65 | 68 | 71
Units on a scale
  Baseline | 99.38 (11.36) | 98.54 (9.51) | 100.53 (12.25) | 100.03 (10.56)
  Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Day 28 | 88.69 (20.18) | 88.94 (17.03) | 85.18 (17.67) | 78.04 (15.78)
Statistical Analysis 1: Comparison: Placebo vs RO6889450 45 mg; Test type: Other; p = 0.849, Mixed Models Analysis; treatment effect = 0.60, 90% CI 2-sided [-4.58 to 5.78]
Statistical Analysis 2: Comparison: Placebo vs RO6889450 150 mg; Test type: Other; p = 0.362, Mixed Models Analysis; treatment effect = -2.83, 90% CI 2-sided [-7.96 to 2.29]
Statistical Analysis 3: Comparison: Placebo vs Risperidone 4 mg; Test type: Other; p = 0.001, Mixed Models Analysis; treatment effect = -10.45, 90% CI 2-sided [-15.46 to -5.43]

2. Secondary Outcome: Change From Baseline in PANSS Factor Scores at Week 4
Description: PANSS factors are modified groupings of the 30 PANSS items from the original three subscales (positive, negative, and general psychopathology). Each item is rated on a scale of 1 (absent) to 7 (most extreme). The positive symptom factor contains 8 items (score range 8-56); the negative symptom and disorganized thought/cognition factors contain 7 items (score range 7-49); the uncontrolled hostility/excitement, expressive deficit, and anxiety/depression factors contain 4 items (score range 4-28); and the avolition domain contains 3 items (score range 3-21). The negative and positive totals each have a range of 7-49 and the general total has a range of 16-112. Higher scores indicate higher symptom severity.
Time Frame: Week 4 (Day 28)
Population: The EAP included all randomized participants who received at least one dose of study medication and who had primary efficacy assessments at baseline and on at least one occasion post-baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 72 | 65 | 68 | 71
Units on a scale
  Anxiety/Depression - Baseline | 11.58 (3.39) | 12.91 (2.92) | 11.54 (3.40) | 12.58 (3.67)
  Anxiety/Depression - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Anxiety/Depression - Day 28 | 9.56 (4.03) | 9.88 (4.15) | 9.06 (4.08) | 8.50 (4.09)
  Avolition - Baseline | 15.99 (3.16) | 15.86 (2.83) | 16.38 (3.25) | 16.20 (2.73)
  Avolition - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Avolition - Day 28 | 14.04 (3.70) | 13.67 (4.42) | 13.73 (3.69) | 12.93 (3.44)
  Disorganized thought/Cognition - Baseline | 21.86 (4.43) | 21.43 (4.66) | 22.50 (4.82) | 21.45 (4.87)
  Disorganized thought/Cognition - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Disorganized thought/Cognition - Day 28 | 19.69 (6.25) | 20.63 (4.94) | 19.41 (6.44) | 17.07 (4.66)
  Expressive deficit - Baseline | 10.89 (3.97) | 10.31 (3.96) | 10.90 (3.79) | 10.23 (3.43)
  Expressive deficit - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Expressive deficit - Day 28 | 10.81 (4.01) | 10.69 (4.39) | 10.16 (4.18) | 10.71 (3.67)
  Totals general - Baseline | 48.42 (6.24) | 48.69 (5.49) | 48.68 (6.57) | 48.89 (6.29)
  Totals general - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Totals general - Day 28 | 42.43 (10.68) | 43.71 (9.06) | 40.43 (8.94) | 37.07 (8.12)
  Negative symptom factor score - Baseline | 23.58 (5.44) | 23.02 (5.19) | 23.81 (5.36) | 23.34 (4.55)
  Negative symptom factor score - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Negative symptom factor score - Day 28 | 21.63 (6.04) | 21.27 (6.63) | 20.80 (5.70) | 20.39 (5.55)
  Totals negative - Baseline | 24.10 (5.29) | 23.65 (4.50) | 24.59 (4.87) | 23.65 (3.78)
  Totals negative - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Totals negative - Day 28 | 22.65 (5.81) | 21.82 (5.85) | 22.53 (5.41) | 21.45 (5.13)
  Positive symptom factor score - Baseline | 31.40 (3.59) | 30.66 (3.84) | 32.03 (4.89) | 31.15 (3.73)
  Positive symptom factor score - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Positive symptom factor score - Day 28 | 27.72 (7.03) | 28.06 (6.14) | 26.63 (7.16) | 24.21 (5.38)
  Totals positive - Baseline | 26.86 (3.60) | 26.20 (4.19) | 27.26 (5.13) | 27.49 (3.95)
  Totals positive - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Totals positive - Day 28 | 23.61 (6.64) | 23.41 (6.14) | 22.22 (6.50) | 19.52 (5.11)
  Uncontrolled hostility/excitement - Baseline | 10.94 (3.94) | 10.52 (4.07) | 10.65 (4.12) | 11.51 (3.90)
  Uncontrolled hostility/excitement - Day 28: number analyzed (Participants) | 54 | 49 | 51 | 56
  Uncontrolled hostility/excitement - Day 28 | 10.09 (4.83) | 9.10 (4.33) | 9.27 (4.22) | 7.86 (4.06)

3. Secondary Outcome: Proportion of Participants With at Least 20% or 50% Improvement From Baseline in the PANSS Total Score
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: Proportion expressed as percentage
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 72 | 65 | 68 | 71
Proportion expressed as percentage
  20% improvement - Week 1 | 18.1 | 26.2 | 27.9 | 25.4
  20% improvement - Week 2 | 26.4 | 24.6 | 36.8 | 43.7
  20% improvement - Week 3 | 31.9 | 32.3 | 38.2 | 59.2
  20% improvement - Week 4 | 30.6 | 32.3 | 36.8 | 59.2
  50% improvement - Week 1 | 0 | 1.5 | 1.5 | 2.8
  50% improvement - Week 2 | 2.8 | 3.1 | 4.4 | 4.2
  50% improvement - Week 3 | 2.8 | 7.7 | 2.9 | 14.1
  50% improvement - Week 4 | 8.3 | 7.7 | 8.8 | 14.1

4. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Scores
Description: The CGI-S measures global severity of illness at a given point in time using a 7-point scale, where 1 = no symptoms and 7 = very severe symptoms.
Time Frame: Week 4 (Day 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 72 | 65 | 68 | 71
Units on a scale
  Baseline | 5.13 (0.50) | 5.09 (0.52) | 5.25 (0.63) | 5.27 (0.61)
  Day 28 | 4.42 (1.07) | 4.35 (0.99) | 4.29 (0.85) | 3.88 (0.94)

5. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Scores
Description: The CGI-I measures change from the baseline state at subsequent visits using a 7-point scale, where 1 = very much improved and 7 = very much worse.
Time Frame: Week 4 (Day 28)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 69 | 60 | 66 | 68
Units on a scale
  Day 7 | 3.87 (0.86) | 3.60 (0.76) | 3.56 (0.88) | 3.40 (0.87)
  Day 14: number analyzed (Participants) | 63 | 59 | 60 | 67
  Day 14 | 3.63 (0.94) | 3.39 (0.95) | 3.33 (0.90) | 2.99 (1.01)
  Day 21: number analyzed (Participants) | 59 | 53 | 55 | 62
  Day 21 | 3.47 (1.19) | 3.28 (1.06) | 3.13 (1.06) | 2.79 (1.01)
  Day 28: number analyzed (Participants) | 52 | 49 | 52 | 56
  Day 28 | 3.27 (1.29) | 3.27 (1.17) | 2.96 (0.93) | 2.43 (0.89)

6. Secondary Outcome: PANSS Total Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo - RO6889450 45 mg | Placebo - RO6889450 150 mg | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 25 | 25 | 41 | 45 | 53
Units on a scale
  Baseline | 103.44 (12.58) | 99.12 (10.16) | 98.66 (9.64) | 99.00 (11.37) | 100.30 (11.49)
  Week 12: number analyzed (Participants) | 10 | 11 | 28 | 20 | 31
  Week 12 | 75.10 (17.53) | 76.73 (21.09) | 76.25 (17.89) | 79.30 (13.68) | 67.74 (11.50)

7. Secondary Outcome: Proportion of Participants With at Least 20% or 50% Improvement in the PANSS Total Score up to Week 12
Description: as for outcome 1
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 2
Measure: Number; unit: Proportion expressed as a percentage
Arm/Group | Placebo - RO6889450 45 mg | Placebo - RO6889450 150 mg | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 25 | 25 | 41 | 45 | 53
Proportion expressed as a percentage
  Week 4 | 40.0 | 36.0 | 46.3 | 53.3 | 75.5
  Week 8 | 36.0 | 28.0 | 43.9 | 37.8 | 69.8
  Week 12 | 28.0 | 28.0 | 48.8 | 28.9 | 50.9

8. Secondary Outcome: CGI-S up to Week 12
Description: as for outcome 4
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo - RO6889450 45 mg | Placebo - RO6889450 150 mg | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 25 | 25 | 41 | 45 | 53
Units on a scale
  Baseline | 5.28 (0.54) | 5.16 (0.47) | 5.05 (0.50) | 5.16 (0.60) | 5.26 (0.62)
  Week 12: number analyzed (Participants) | 9 | 11 | 27 | 20 | 31
  Week 12 | 3.33 (1.00) | 3.73 (1.27) | 3.56 (1.01) | 3.90 (0.85) | 3.06 (0.81)

9. Secondary Outcome: CGI-I up to Week 12
Description: as for outcome 5
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo - RO6889450 45 mg | Placebo - RO6889450 150 mg | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 25 | 25 | 41 | 45 | 53
Units on a scale
  Day 7: number analyzed (Participants) | 24 | 25 | 41 | 45 | 53
  Day 7 | 3.54 (0.66) | 3.76 (0.78) | 3.54 (0.78) | 3.56 (0.84) | 3.38 (0.84)
  Week 12: number analyzed (Participants) | 9 | 11 | 27 | 20 | 31
  Week 12 | 2.33 (1.00) | 2.73 (1.56) | 2.30 (0.91) | 2.65 (0.93) | 2.00 (0.82)

10. Secondary Outcome: Participants Ready for Discharge From First Randomized Treatment Intake to Readiness for Discharge as Assessed by the Readiness for Discharge Questionnaire (RDQ) at 4-Week Treatment
Description: The RDQ is a tool used to assess inpatients with schizophrenia on their readiness for discharge from inpatient treatment. It consists of five items that assess suicidality/homicidality, control of aggression/impulsivity, activities of daily living, medication-taking, and delusions/hallucinations interfering with functioning and global status. An additional item examines the overall clinical state of the patient and the final question assesses readiness for discharge. The values reported are the proportion (expressed as a percentage) of participants in each analysis group considered ready for discharge according to the RDQ.
Time Frame: after 4-week treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | RO6889450 45 mg | RO6889450 150 mg | Risperidone 4 mg
Number analyzed (Participants) | 64 | 54 | 61 | 69
Percentage of participants | 88.9 [79.3 to 95.1] | 83.1 [71.7 to 91.2] | 89.7 [79.9 to 95.8] | 97.2 [90.2 to 99.7]

11. Secondary Outcome: Plasma Concentration of RO6889450
Time Frame: Day 7 - Day 336
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo - RO6889450 45 mg | Placebo - RO6889450 150 mg | RO6889450 45 mg | RO6889450 150 mg
Number analyzed (Participants) | 25 | 25 | 71 | 69
ng/mL
  Day 7: number analyzed (Participants) | 0 | 0 | 57 | 65
  Day 7 |  |  | 99.50 (69.2) | 423.83 (43.2)
  Day 14: number analyzed (Participants) | 0 | 0 | 58 | 59
  Day 14 |  |  | 91.53 (111.4) | 463.21 (73.6)
  Day 28: number analyzed (Participants) | 5 | 4 | 45 | 47
  Day 28 | 49.67 (155.4) | 212.27 (25.0) | 94.57 (108.1) | 419.41 (93.0)
  Day 42: number analyzed (Participants) | 13 | 15 | 35 | 36
  Day 42 | 59.99 (248.3) | 274.58 (208.8) | 108.57 (76.4) | 390.65 (138.4)
  Day 56: number analyzed (Participants) | 10 | 12 | 33 | 31
  Day 56 | 70.99 (320.4) | 217.65 (491.6) | 108.59 (55.5) | 237.42 (541.2)
  Day 84: number analyzed (Participants) | 12 | 12 | 33 | 31
  Day 84 | 77.11 (85.5) | 165.99 (963.0) | 92.24 (128.5) | 265.09 (353.6)
  Day 168: number analyzed (Participants) | 0 | 0 | 2 | 2
  Day 168 |  |  | 95.39 (46.0) | 733.98 (65.5)
  Day 336: number analyzed (Participants) | 0 | 0 | 1 | 2
  Day 336 |  |  | 4.13 (NA) — The value was not estimable for data from a single participant. | 139.71 (120.6)

ADVERSE EVENTS:
Time Frame: 4 weeks for double-blind treatment period Up to 48 weeks for extension period
Groups:
- RO6889450 45 mg (Double-blind Treatment Period); RO6889450 45 mg (Extension Period): Participants received 45 mg of RO6889450 QD for 4, 12, or 48 weeks.
- RO6889450 150 mg (Double-blind Treatment Period); RO6889450 150 mg (Extension Period): Participants received 150 mg of RO6889450 QD for 4, 12, or 48 weeks.
- Risperidone 4 mg (Double-blind Treatment Period); Risperidone 4 mg (Extension Period): Participants received 4 mg of risperidone QD for 4, 12, or 48 weeks.
Arm/Group | Placebo | RO6889450 45 mg (Double-blind Treatment Period) | RO6889450 150 mg (Double-blind Treatment Period) | Risperidone 4 mg (Double-blind Treatment Period) | Placebo - RO6889450 45 mg | Placebo - RO6889450 150 mg | RO6889450 45 mg (Extension Period) | RO6889450 150 mg (Extension Period) | Risperidone 4 mg (Extension Period)
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/65 | 0/68 | 0/71 | 0/25 | 1/25 | 0/41 | 0/45 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/72 | 2/65 | 1/68 | 0/71 | 3/25 | 3/25 | 1/41 | 6/45 | 1/53
Other Adverse Events (participants affected / at risk) | 23/72 | 14/65 | 23/68 | 36/71 | 5/25 | 6/25 | 7/41 | 12/45 | 5/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | RO6889450 45 mg (Double-blind Treatment Period) (N=65) | RO6889450 150 mg (Double-blind Treatment Period) (N=68) | Risperidone 4 mg (Double-blind Treatment Period) (N=71) | Placebo - RO6889450 45 mg (N=25) | Placebo - RO6889450 150 mg (N=25) | RO6889450 45 mg (Extension Period) (N=41) | RO6889450 150 mg (Extension Period) (N=45) | Risperidone 4 mg (Extension Period) (N=53)
Schizophrenia (Psychiatric disorders) | 1 | 2 | 0 | 0 | 3 | 2 | 1 | 5 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | RO6889450 45 mg (Double-blind Treatment Period) (N=65) | RO6889450 150 mg (Double-blind Treatment Period) (N=68) | Risperidone 4 mg (Double-blind Treatment Period) (N=71) | Placebo - RO6889450 45 mg (N=25) | Placebo - RO6889450 150 mg (N=25) | RO6889450 45 mg (Extension Period) (N=41) | RO6889450 150 mg (Extension Period) (N=45) | Risperidone 4 mg (Extension Period) (N=53)
Anxiety (Psychiatric disorders) | 6 | 3 | 2 | 5 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 5 | 5 | 0 | 0 | 1 | 1 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 8 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 4 | 5 | 6 | 0 | 0 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 6 | 0 | 1 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 5 | 0 | 0 | 1 | 1 | 0
Weight increased (Investigations) | 1 | 2 | 0 | 8 | 1 | 1 | 0 | 1 | 4
Schizophrenia (Psychiatric disorders) | 3 | 2 | 0 | 1 | 4 | 3 | 2 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT04512066/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT04512066/SAP_001.pdf